CLINICAL TRIAL: NCT01526811
Title: Post-market Study on Endurant™ Stent Graft System in the Treatment of Infra-renal Abdominal Aortic Aneurysms
Brief Title: Endurant™ Stent Graft System in the Treatment of Infra-renal Abdominal Aortic Aneurysms (ENDURANT France)
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: P#8888
Record Dates: First submitted 2012-01-27; First posted 2012-02-06 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Aneurysm; Aortic Aneurysm; Aortic Aneurysm, Abdominal; Vascular Diseases; Cardiovascular Diseases; Aortic Diseases
Keywords: Endurant; Stent Graft; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aneurysm; Aortic Aneurysm; Aortic Aneurysm, Abdominal; Vascular Diseases; Cardiovascular Diseases; Aortic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AAA patients: Subjects presenting with a non-ruptured infra-renal abdominal aortic aneurysm (AAA) and requiring endovascular treatment with Endurant™ Stent Graft, and who meet the inclusion/exclusion criteria are intended to participate in this non-interventional study
  Interventions: Device: Endurant Stent graft

INTERVENTIONS:
Device: Endurant Stent graft — Endurant Stent graft implantation
  Other Names: EVAR

SUMMARY:
The purpose of this study is to assess the benefits of endovascular repair with Endurant Stent Graft System by documenting overall mortality, complications, the rate of conversion to open surgical repair, and the development and rupture of the aneurysm on a long term, i.e. at 5 years, in a cohort of patients representative of the population treated under real-life conditions of use in France.

DETAILED DESCRIPTION:
Data regarding the use under routine practice of abdominal aortic stent grafts in France are expected by the French National Authority for Health (HAS). Therefore, in its opinion report from July 13, 2010, HAS makes the maintenance of reimbursement approval of each stent graft dependent on the presentation of results of a specific follow-up study carried out in a cohort of patients representative of the French population treated under real-life conditions of use. This prospective cohort study must involve at least 150 patients implanted after registration on the LPPR (List of Products and Services qualifying for Reimbursement). The results of the follow-up study must be forwarded to the National Committee for Evaluation of Medical Devices and Health Technologies (CNEDiMTS) for examination once a year. The assessment of this follow-up could lead to the recommendation by CNEDiMTS to continue or stop the reimbursement of the concerned stent graft.

In France, The Endurant™ Stent Graft System is registered on the LPPR for a period of 3 years since September 13, 2011. In order to comply with HAS expectations, Medtronic Bakken Research Center is setting up this long term non-interventional study on the Endurant stent graft.

ELIGIBILITY:
Inclusion Criteria:

* Patient with age ≥18 years, who is able to understand the information given by the investigator regarding the collection and release of his/her personal information and who is able to oppose to this collection and release.
* Any patient requiring placement of an abdominal aortic stent graft for the treatment of a non-ruptured infra-renal abdominal aortic aneurysm.
* Patient not opposed to the collection and release of his/her personal information
* Intention of physician to implant electively the Endurant™ Stent Graft System

Exclusion Criteria:

* Patient in whom clinical follow-up will not be possible i.e. patient not able to come back for follow-up visits (ex. patient living abroad)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with a non-ruptured infra-renal abdominal aortic aneurysm (AAA) and requiring endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-03; Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | through 5 years
Aneurysm diameter's change | through 5 years
Stent graft endoleaks (type I, II and III) | through 5 years
Stent Graft migration | through 5 years
Conversion to open surgical repair | through 5 years
Surgical or endovascular secondary procedures | through 5 years
Aneurysm-related mortality | through 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Becquemin, MD, PhD, Principal Investigator — Groupe Hospitalier Henri-Mondor, Créteil, France
Locations (20):
- France (20):
  - Centre Hospitalier d'Avignon, Avignon
  - CHU de Besancon, Hôpital Jean Minjoz, Besançon
  - Médipôle de Savoie, Challes-les-Eaux
  - Hôpital Privé Sainte Marie, Chalon-sur-Saône
  - Groupe Hospitalier Henri-Mondor, Créteil
  - Clinique Claude Bernard, Ermont
  - Clinique du Mousseau, Évry
  - Clinique de la Présentation, Fleury-les-Aubrais
  - CHU Limoges, Limoges
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Paul Desbief, Marseille
  - Hôpital Ambroise Paré, Marseille
  - Hôpital Saint Joseph, Marseille
  - Clinique du Millenaire, Montpellier
  - CHU Nice, Hôpital Saint-Roch, Nice
  - Polyclinique Quimper Sud, Quimper
  - Clinique Belledonne, Saint-Martin-d'Hères
  - CHl Toulon - La Seyne sur Mer, Toulon
  - Clinique Sarrus Teinturiers, Toulouse
  - Clinique Saint Joseph, Trélazé